CLINICAL TRIAL: NCT04813939
Title: Is Bio-adrenomedullin (Bio-ADM) a Prognostic Factor in Patients With COVID-19 Treated in the ICU?
Status: Terminated | Type: Observational
Why Stopped: Enrollment was terminated because of the poor recruitment rate.
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: 042021
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: bio-adrenomedullin; point of care; sepsis
MeSH Terms: conditions — COVID-19; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: IB10 sphingotest® bio-ADM® apparatus (Sphingotec GmbH, Hennigsdorf, Germany) — Point of care assessment of bio-adrenomedullin concentration will be performed using the IB10 sphingotest® bio-ADM® apparatus (Sphingotec GmbH, Hennigsdorf, Germany) on the 1,3,5-day ICU stay in COVID-19 patients. The method used is a double monoclonal sandwich immunoassay to measure the concentration of C-terminal amidated, biologically active adrenomedullin (bio-ADM) in whole blood. Additional measurement of bio-ADM will be performed as standard monitoring in patients suspected of septic complications of the course of COVID-19.

SUMMARY:
This is prospective, observational study using point of care test to determine bio-ADM whole blood concentrations and its predictive value in patients with COVID-19 treated in the ICU.

DETAILED DESCRIPTION:
About 5% of all patients infected with the SARS-CoV-2 virus require treatment in the ICU. The main reason for admission to the ICU is acute hypoxemic respiratory failure, which in most cases is associated with the need for mechanical ventilation. The progression of lung damage affects not only alveoli but also endothelium of the pulmonary vessels. Occurring endotheliopathy is caused by direct infection with SARS-CoV-2 virus and activation of the immune system leading to an increased inflammatory reaction. Damage to the endothelium barrier with concomitant cytokine storm lead to activation of the coagulation system and formation of microthrombotic events in the vascular bed, resulting in thromboembolic complications and development of multiorgan failure. The reflection of the above pathophysiological phenomena in laboratory tests is a significant increase in the concentration of D-dimers. At present, no specific markers of endotheliopathy in patients with SARS-CoV-2 are known.

Adrenomedullin (ADM) is a peptide hormone that plays a key role in regulating the function of the endothelium, by modulating its integrity and permeability, it also has an effect on the vascular muscle, leading to vasodilation. Recently, the role of ADM has been intensively studied, including in sepsis. Several studies have confirmed an association between elevated ADM levels and poor prognosis in sepsis and septic shock. In these studies, measurements of various adrenomedullin precursors and free, biologically active adrenomedullin (bio-adrenomedullin, bio-ADM) were performed. The role of bio-ADM in the course of COVID -19 remains unclear.

The aim of the study is to determine the baseline concentration of bio-ADM and to determine the dynamic of the concentration changes in three measurements in patients with COVID-19 during ICU treatment. Additional measurement of bio-ADM will be performed as standard monitoring in patients suspected of septic complications of the course of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* polymerase chain reaction (PCR) confirmed COVID-19
* severe stage of pneumonia caused by SARS-CoV-2 requiring oxygen therapy
* informed consent to participate in the study

Exclusion Criteria:

* qualification to palliative care
* life expectancy < 48 h
* mechanical ventilation at the beginning of the hospitalization
* transfer from other ICU
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients from emergency department and intermediate department meeting the eligibility criteria will be enrolled to the study.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 28-days
  28-day mortality will be assessed

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) Score and its changes over time | 28-days
  Occurrence of multiorgan failure expressed in SOFA scores
Need for catecholamines | 28-days
  Need for catecholamines (drug, highest/lowest dose, duration)
Need for renal replacement therapy | 28-days
  Need for renal replacement therapy (duration)
Need for mechanical ventilation | 28-days
  Need for mechanical ventilation (duration)
Changes of partial pressure of oxygen in arterial blood (PaO2) / fraction of inspired oxygen (FiO2) during treatment in ICU | 28-days
  PaO2/FiO2
Changes in D-dimer | 28-days
  Changes in D-dimer (in ng/ml)
Changes in blood lactate levels | 28-days
  Changes in blood lactate levels (in mg/dl)
Changes C reactive protein (CRP) | 28-days
  Changes CRP (in mg/l)
Changes in procalcitonin levels | 28-days
  Changes in procalcitonin levels (in ng/ml)
Changes in creatinine levels | 28-days
  Changes in creatinine levels (in mg/dl)

OTHER OUTCOMES:
Sepsis complicating the course of COVID-19 during ICU treatment | 28-days
  Occurrence of sepsis complicating the course of COVID-19 during ICU treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Zatorski, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No